CLINICAL TRIAL: NCT00412438
Title: Investigation of Genetic Risk of Atrial Fibrillation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Nagoya University (Other)
Other Study IDs: RIEM-G-1
Record Dates: First submitted 2006-12-15; First posted 2006-12-18 (Estimated); Last update posted 2006-12-18 (Estimated); Status verified 2006-12

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other

SUMMARY:
The atrial fibrillation (AF) is the most common cardiac rhythm disturbance that is responsible for substantial morbidity and mortality independent of associated heart disease or other risk factors. Even in the absence of preexisting cardiovascular disease, AF remains significantly associated with excess mortality rates. The current unsatisfactory treatment for AF comes from lack of understanding of the pathophysiology of AF. The purpose of this study is to identify gene polymorphisms that confer susceptibility to atrial fibrillation. Patients with AF（N=500） and healthy volunteer（N=1000） without AF are enrolled in this study. Patients with coronary artery disease, severe valvular heart disease, cardiomyopathy or heart failure were excluded from the study.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of atrial fibirillation

Exclusion Criteria:

* coronary artery disease
* severe valvular heart disease
* cardiomyopathy
* heart failure

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1000
Dates: Start 2006-10

CONTACTS AND LOCATIONS:
Overall Officials: Kenji Yasui, MD, Phd, Study Chair — Department of Bio-information Analysis, Research Institute of Enviromental Medicine, Nagoya University
Locations (1):
- Department of Bio-information Analysis, Research Institute of Enviromental Medicine, Nagoya University, Nagoya, Aichi-ken, Japan